CLINICAL TRIAL: NCT05794048
Title: METabolic PROFILE of Hepatocarcinoma and Pancreatic Tumors
Acronym: PROMETHEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP210017
Record Dates: First submitted 2022-10-17; First posted 2023-03-31 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Hepatocarcinoma; Pancreatic Tumor
Keywords: Hepatocarcinoma; Pancreatic Tumor
MeSH Terms: conditions — Carcinoma, Hepatocellular; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hepatocellular carcinoma (Experimental): Patients with hepatocellular carcinoma
  Interventions: Biological: Hepatocellular carcinoma
- Pancreatic adenocarcinoma (Experimental): Patients with pancreatic adenocarcinoma
  Interventions: Biological: Pancreatic adenocarcinoma
- Pancreatic neuroendocrine tumor (Experimental): Patients with pancreatic neuroendocrine tumor
  Interventions: Biological: Pancreatic neuroendocrine tumor

INTERVENTIONS:
Biological: Hepatocellular carcinoma — Tumor and liver biopsy
  Arms: Hepatocellular carcinoma
Biological: Pancreatic adenocarcinoma — Tumor and pancreatic biopsy
  Arms: Pancreatic adenocarcinoma
Biological: Pancreatic neuroendocrine tumor — Tumor and pancreatic biopsy
  Arms: Pancreatic neuroendocrine tumor

SUMMARY:
Hepatic (hepatocellular carcinoma (HCC)) and pancreatic (pancreatic adenocarcinoma (ADKP); pancreatic neuroendocrine tumors (TNEP)) primary tumors are the most common malignant tumors of the hepato-bilio-pancreatic system and represent a major public health issue. At present, the management of these tumors is based on recommendations based on the existence of rudimentary prognostic and theranostics markers that do not sufficiently accurately reflect the heterogeneity of tumor biology. It therefore seems essential to identify new and more relevant markers in order to optimize the care of these patients in daily practice.

Metabolic reprogramming is now recognized as an essential feature of cancer cells, allowing them to fuel and maintain their proliferation and tumor growth. Such metabolic reprogramming requires modification of several energy pathways, the most commonly recognized being the transition from energy metabolism based on oxidative phosphorylation to energy metabolism based on glycolysis, even under aerobic conditions (Warburg effect). In this context, the investigators hypothesized that the consumption of nutrients by the tumor cell differs significantly from that of the normal cell in order to support its increased energy needs, and that this important and specific metabolic reprogramming would be correlated with the histo-prognostic and theranostics factors of these tumors. Preliminary analyses on surgical resection parts conducted by the various partners in 2019 made it possible to characterize the metabolic signatures of a series of HCC and ADKP resected using the Metafora biosystems technology platform. These signatures reflect a metabolic program characteristic of these tumors, which reveal strong specificities. Similarly, a candidate signature correlating with the presence of vascular microscopic invasion has been identified in HCC, and the level of activation of glycolysis and glutaminolysis by certain ADKP cells also appears as a trait of interest vis-à-vis the aggressiveness of this cancer.

Thus, the current project will aim to confirm the feasibility of identifying specific prognostic and theranostics metabolic signatures early, on biopsy samples and / or circulating blood cells.

DETAILED DESCRIPTION:
Primary liver tumours (hepatocellular carcinoma (HCC)) and pancreatic tumours (pancreatic adenocarcinoma (ADKP); pancreatic neuroendocrine tumours (NETs)) are the most frequent malignant tumours of the hepatobiliopancreatic system and represent a major public health issue. One of the main lines of research for these tumors consists in the early identification of prognostic and theranostic factors to adapt the management of patients as closely as possible to the specificities of their pathology. This identification is currently sorely lacking in daily clinical practice. Thus, unlike what is done for other types of neoplastic pathologies such as breast cancer, the management of primary liver and pancreatic tumors is still often based on recommendations based on the existence of rudimentary prognostic and theranostic markers that do not reflect sufficiently faithfully the heterogeneity of tumor biology. It is therefore essential to identify new, more relevant markers in order to optimize the management of these patients in daily practice.

Metabolic reprogramming is now recognized as an essential characteristic of cancer cells, allowing them to fuel and maintain their proliferation and tumor growth. Such metabolic reprogramming requires modification of several energy pathways, the most commonly recognized being the shift from energy metabolism based on oxidative phosphorylation to energy metabolism based on glycolysis, even under aerobic conditions (Warburg effect). Other metabolic pathways such as increased glutaminolysis have recently been identified. In this context, we hypothesized that the consumption of nutrients by the tumor cell differs significantly from that of the normal cell in order to support its increased energy needs, and that this important and specific metabolic reprogramming would be correlated with the histo-prognostic and theranostic factors of these tumors. Within ADKPs, 2 molecular subtypes have been described: a very aggressive, "basal-like" subtype with increased glycolytic metabolism and metastatic properties and a "classical" subtype, better differentiated with better prognosis. The identification of these subtypes is currently only possible by RNA-seq, a technology not practiced routinely. Similarly, metabolism appears to define a subgroup of aggressive NETs. Indeed, NETs with high glucose uptake, visible on 18FDG PET-CT scan, have a worse prognosis. This type of examination also showed that there was spatial metabolic heterogeneity (primary tumor vs. metastasis) and temporal metabolic heterogeneity in these tumors and that the latter was correlated with prognosis.

Preliminary analyses conducted by the various partners in 2019 made it possible to characterize the metabolic signatures of a series of resected HCC and ADKP using Metafora biosystems' technological platform.

These signatures reflect a metabolic program characteristic of these tumors, which reveal strong specificities. Similarly, a candidate signature correlating with the presence of microscopic vascular invasion has been identified in HCC, and the level of activation of glycolysis and glutaminolysis by some ADKP cells also appears as a trait of interest vis-à-vis the aggressiveness of this cancer.

As these results were obtained on surgical resection parts, the current project will therefore aim to confirm the feasibility of identifying specific prognostic and theranostic metabolic signatures early, on biopsy sampling or circulating blood cells.

This multicenter study includes 300 patients (100 patients for each tumor type) and aims to identify a prognostic metabolic signature from tumor tissue samples of HCC, ADKP and pancreatic NETs.

ELIGIBILITY:
Inclusion criteria :

Common criteria:

* Patient aged 18 or over
* Informed and having signed the consent to participate
* Affiliated with a social security scheme or entitled

  1- Patients with hepatocellular carcinoma
* Having a HCC eligible for surgical treatment (liver resection or liver transplantation) not requiring preoperative anti-tumor treatment as validated by the multidisciplinary consultation meeting for primary hepatic tumors
* OR having a HCC not eligible for curative treatment (liver resection, liver transplantation, tumor ablation), as validated by the multidisciplinary consultation meeting for primary hepatic tumors 2- Patients with pancreatic adenocarcinoma or pancreatic neuroendocrine tumor
* Having ADKP or NET eligible for surgical treatment (duodenopancreatectomy, left pancreatectomy, enucleation, central pancreatectomy, hepatic metastasectomy) with or without preoperative anti-tumor treatment as validated by the multidisciplinary consultation meeting.
* OR with an unresectable ADKP or TNEP, with only medical treatment plan as validated by the multidisciplinary consultation meeting

Exclusion criteria :

Criteria common to all patients:

* Pregnancy and lactation
* Lack of informed, written and signed consent
* Adult person subject to a legal protection measure or unable to express consent
* Patient under State Medical Aid (AME)
* Person deprived of liberty by a judicial or administrative decision
* Person undergoing psychiatric care

  1- Patients with hepatocellular carcinoma
* Suspicion of mixed tumor (hepatocholangiocarcinoma) or intrahepatic cholangiocarcinoma
* History of systemic or locoregional anti-tumor treatment in the target tumor
* Contraindication to a liver biopsy
* Decompensated cirrhosis 2- Patients with pancreatic adenocarcinoma or pancreatic neuroendocrine tumor
* Suspicion of mixed tumor (MINEN) or intra-pancreatic cholangiocarcinoma
* Contraindication to a pancreatic / hepatic biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2026-09-08 (Estimated)

PRIMARY OUTCOMES:
Prognostic metabolic signatures of HCC | 24 months
  Identify prognostic metabolic signatures obtained from operative specimens and biopsies of hepatocellular carcinoma (HCC).
  As this is an exploratory pilot study, it does not include primary and secondary endpoints. Metabolic signatures will be statistically processed to correlate with clinical prognosis.
Prognostic metabolic signatures of ADKP | 36 months
  Identify prognostic metabolic signatures obtained from operative specimens and biopsies of pancreatic adenocarcinoma (ADKP).
  As this is an exploratory pilot study, it does not include primary and secondary endpoints. Metabolic signatures will be statistically processed to correlate with clinical prognosis.
Prognostic metabolic signatures of TNEP. | 24 months
  Identify prognostic metabolic signatures obtained from operative specimens and biopsies of pancreatic neuroendocrine tumors (TNEP).
  As this is an exploratory pilot study, it does not include primary and secondary endpoints. Metabolic signatures will be statistically processed to correlate with clinical prognosis.
Theranostic metabolic signatures of HCC. | 24 months
  Identify theranostic metabolic signatures obtained from operative specimens and biopsies of hepatocellular carcinoma (HCC).
  As this is an exploratory pilot study, it does not include primary and secondary endpoints. Metabolic signatures will be statistically processed to correlate with clinical prognosis.
Theranostic metabolic signatures of ADKP. | 36 months
  Identify theranostic metabolic signatures obtained from operative specimens and biopsies of pancreatic adenocarcinoma (ADKP).
  As this is an exploratory pilot study, it does not include primary and secondary endpoints. Metabolic signatures will be statistically processed to correlate with clinical prognosis.
Theranostic metabolic signatures of TNEP. | 24 months
  Identify theranostic metabolic signatures obtained from operative specimens and biopsies of pancreatic neuroendocrine tumors (TNEP).
  As this is an exploratory pilot study, it does not include primary and secondary endpoints. Metabolic signatures will be statistically processed to correlate with clinical prognosis.

SECONDARY OUTCOMES:
Identification of circulating HCC tumor cells based on detection of their metabolic profile | 24 months
  As this is a pilot study, these metabolic signatures will then be statistically processed to correlate them with clinical prognosis; This is not an evaluation criterion stricto sensu.
Identification of circulating ADKP tumor cells based on detection of their metabolic profile | 24 months
  As this is a pilot study, these metabolic signatures will then be statistically processed to correlate them with clinical prognosis; This is not an evaluation criterion stricto sensu.
Identification of circulating TNEP tumor cells based on detection of their metabolic profile | 36 months
  As this is a pilot study, these metabolic signatures will then be statistically processed to correlate them with clinical prognosis; This is not an evaluation criterion stricto sensu.
Comparison of circulating tumor cells with detection based solely on an epithelial marker | 36 months
  As this is a pilot study, these metabolic signatures will then be statistically processed to correlate them with clinical prognosis; This is not an evaluation criterion stricto sensu.
Identification of prognostic metabolic signatures obtained on circulating tumor cells of HCC. | 24 months
  As this is a pilot study, these metabolic signatures will then be statistically processed to correlate them with clinical prognosis; This is not an evaluation criterion stricto sensu.
Identification of prognostic metabolic signatures obtained on circulating tumor cells of ADKP | 24 months
  As this is a pilot study, these metabolic signatures will then be statistically processed to correlate them with clinical prognosis; This is not an evaluation criterion stricto sensu.
Identification of prognostic metabolic signatures, obtained on circulating tumor cells of TNEP | 36 months
  As this is a pilot study, these metabolic signatures will then be statistically processed to correlate them with clinical prognosis; This is not an evaluation criterion stricto sensu.
Identification of theranostic metabolic signatures obtained on circulating tumor cells of HCC | 24 months
  As this is a pilot study, these metabolic signatures will then be statistically processed to correlate them with clinical prognosis; This is not an evaluation criterion stricto sensu.
Identification of theranostic metabolic signatures, obtained on circulating tumor cells of ADKP | 24 months
  As this is a pilot study, these metabolic signatures will then be statistically processed to correlate them with clinical prognosis; This is not an evaluation criterion stricto sensu.
Identification of theranostic metabolic signatures, obtained on circulating tumor cells of TNEP | 36 months
  As this is a pilot study, these metabolic signatures will then be statistically processed to correlate them with clinical prognosis; This is not an evaluation criterion stricto sensu.
Identification of the metabolic profile of blood immune cells. | 36 months
  As this is a pilot study, these metabolic signatures will then be statistically processed to correlate them with clinical prognosis; This is not an evaluation criterion stricto sensu.
Study of prognostic value of metabolic profile of blood immune cells. | 36 months
  As this is a pilot study, these metabolic signatures will then be statistically processed to correlate them with clinical prognosis; This is not an evaluation criterion stricto sensu.
Study of theranostic value of metabolic profile of blood immune cells. | 36 months
  As this is a pilot study, these metabolic signatures will then be statistically processed to correlate them with clinical prognosis; This is not an evaluation criterion stricto sensu.
Comparison of metabolic profiles on biopsy sample. | 36 months
  As this is a pilot study, these metabolic signatures will then be statistically processed to correlate them with clinical prognosis; This is not an evaluation criterion stricto sensu.
Comparison of metabolic profiles on surgical specimen | 36 months
  As this is a pilot study, these metabolic signatures will then be statistically processed to correlate them with clinical prognosis; This is not an evaluation criterion stricto sensu.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Paradis, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Beaujon, Clichy, France